CLINICAL TRIAL: NCT02227329
Title: Prophylactic Ethanol Lock Therapy (ELT) in Patients on Home Parenteral Nutrition: A Prospective Randomized Control Trial.
Brief Title: Prophylactic Ethanol Lock Therapy (ELT) in Patients on Home Parenteral Nutrition
Acronym: ELT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Publication of guidelines advising against the use of ethanol locks.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13-007793
Record Dates: First submitted 2014-08-15; First posted 2014-08-28 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Catheter-related Bloodstream Infection (CRBSI) Nos; Bloodstream Infection Due to Central Venous Catheter; Bloodstream Infection Due to Hickman Catheter
Keywords: Home Parenteral Nutrition; Infection Prevention; CRBSI; Ethanol Lock Therapy
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Ethanol; Vascular Access Devices; Heparin; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ethanol Lock and Normal Saline (Experimental): All patients randomized to the ELT group will receive 3ml of 70% ethanol and saline flush.
  Interventions: Drug: Ethanol; Drug: Normal Saline
- Heparin and Normal Saline (Active Comparator): All patients randomized to this group will receive Heparin lock + saline infusion (current standard of care).
  Interventions: Drug: Heparin Lock; Drug: Normal Saline

INTERVENTIONS:
Drug: Ethanol — Prophylactic ELT will be administered at the time when the HPN is not being infused.
  Other Names: Alcohol lock; Ethanol (EtOH); ELT therapy
  Arms: Ethanol Lock and Normal Saline
Drug: Heparin Lock — 3 mL of 100 U/ml heparin
  Other Names: Hep-Lock; Heparin
  Arms: Heparin and Normal Saline
Drug: Normal Saline
  Other Names: N Saline; 0.9 N saline

SUMMARY:
This study is being implemented to identify the role of prophylactic use of ethanol lock in adult patients on home parenteral nutrition (HPN). Central catheter related blood stream infection is a major complication in patients on HPN. The investigators hypothesize that the prophylactic use of ELT will decrease the number of catheter related blood stream infections compared to the control group. The investigators further hypothesize that with the introduction of prophylactic ELT, the number of infections will decrease.

DETAILED DESCRIPTION:
Catheter-related bloodstream infection (CRBSI) is a serious complication for home parenteral nutrition (HPN) patients causing morbidity, mortality, and prolonged hospitalization. CRBSIs may also result in the need for central venous catheter (CVC) removal and replacement. Current literature supports the use of antibiotics locks in patients with repeated CRBSI. There is a growing concern about the increased risk of microbial resistance with the long term use antibiotic locks. Ethanol lock therapy (ELT) has broad spectrum coverage and includes gram negative bacteria, gram positive bacteria, atypical bacteria, and fungi. Compared with antibiotic and other solution locks, which have limitations, ELT has excellent broad-spectrum bactericidal and fungicidal killing action and poses no problems with development of resistance over time. There is a lack of a randomized controlled study to characterize the role of ELT in adult patients on HPN.

ELIGIBILITY:
Inclusion Criteria:

* Newly started on Home parenteral Nutrition and anticipated duration >3 months.
* Not previously on Home Parenteral Nutrition.
* Providing consent.
* Patients with non-medicare insurance.
* Patients with medicare insurance and a supplementary insurance.
* Patients with single lumen Hickman® catheters.
* No known alcohol addiction.

Exclusion Criteria:

* Failure to provide consent
* Patients with medicare insurance and no other supplemental private insurance
* Patients with a catheter type other than a single lumen Hickman®
* Patients who are on HPN for less than three months
* Pregnant patients
* Patients who have previous proven addiction and dependence to alcohol.
* Patients lacking capacity to provide consent
* Patients who are not be managed by HPN team at investigator's institution

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Salonen BR, Bonnes SL, Vallumsetla N, Varayil JE, Mundi MS, Hurt RT. A prospective double blind randomized controlled study on the use of ethanol locks in HPN patients. Clin Nutr. 2018 Aug;37(4):1181-1185. doi: 10.1016/j.clnu.2017.05.009. Epub 2017 May 17. PMID 28576557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This clinical trial was carried out from July 2014 to April 2016 at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 39 subjects were consented, but one subject was excluded after enrollment due to incompatibility with ongoing treatment (ongoing metronidazole use).
Groups:
- Heparin and Normal Saline: All patients randomized to this group will receive Heparin lock (3 mL of 100 U/ml heparin) + saline infusion (current standard of care).
Period: Overall Study
Arm/Group | Ethanol Lock and Normal Saline | Heparin and Normal Saline
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ethanol Lock and Normal Saline | Heparin and Normal Saline | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16) | 52 (16) | 51 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Catheter-Related Blood Stream Infections
Description: The most common complication in parenteral nutrition is catheter-related blood stream infection (CRBSI), which can lean to increased morbidity, mortality, and prolonged hospitalizations. CRBSI was defined as bacteremia or fungemia in a patient who had an intravascular device and >1 positive blood culture result obtained from the peripheral vein, clinical manifestations of infection (e.g., fever, chills, and/or hypotension), and no apparent source for blood stream infection other than the central venous catheter.
Time Frame: 1 year
Measure: Number; unit: infections
Arm/Group | Ethanol Lock and Normal Saline | Heparin and Normal Saline
Number analyzed (Participants) | 18 | 20
infections | 4 | 1
Statistical Analysis 1: Comparison: Ethanol Lock and Normal Saline vs Heparin and Normal Saline; Test type: Superiority; p = 0.17, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ethanol Lock and Normal Saline | Heparin and Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 4/18 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethanol Lock and Normal Saline (N=18) | Heparin and Normal Saline (N=20)
Catheter-related bloodstream infection (Infections and infestations) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines on chronic intestinal failure in adults advising against ELT, we conducted an interim analysis. The study was terminated early; further study would not change outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes